ATP Level and Cough Sensitivity to ATP in Subjects with Refractory/Unexplained Chronic Cough

NCT05265871

**April 25, 2025** 

**Statistical Analysis Plan** 

IBM SPSS Statistics version 26 was used for analysis. Concentrations of ATP and capsaicin were log-transformed (Lg) for calculation. Normal distribution data was presented as mean±standard deviation, while median (interquartile range) for skewed data. Data were compared by independent-samples t test, Mann-whitney U test or chi-square test. Correlation analysis was conducted using Pearson correlation coefficient. A P value < 0.05 was considered statistically significant.